CLINICAL TRIAL: NCT01096095
Title: Phenylbutyrate in SCA3: a Double-blind, Placebo-controlled Study to Determine Safety and Efficacy of Sodium Phenylbutyrate in Patients With SCA3
Brief Title: Pilot Study of Safety and Efficacy of Sodium Phenylbutyrate in Spinocerebellar Ataxia Type 3
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Regulatory authorities did not allow the entrance of the study drug in the country
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CONEP CAAE 0527.0.001.000-07
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2010-05

CONDITIONS: Spinocerebellar Ataxia Type 3
Keywords: SCA; Spinocerebellar Ataxia; Sodium Phenylbutyrate; Machado-Joseph Disease; Treatment
MeSH Terms: conditions — Machado-Joseph Disease; Spinocerebellar Ataxias | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Sodium phenylbutyrate (Experimental): Active drug
  Interventions: Drug: Sodium Phenylbutyrate

INTERVENTIONS:
Drug: Placebo — Powdered placebo in sachets containing each 3g. At the start of the study, the dose will be 15g/day (five sachets).
  Arms: Placebo
Drug: Sodium Phenylbutyrate — Powdered sodium phenylbutyrate in sachets containing each 3g. At the start of the study, the dose will be 15g/day (five sachets) and may be reduced in case of mild adverse events.
  Arms: Sodium phenylbutyrate

SUMMARY:
DESIGN: Pilot, Phase II, double-blind, placebo-controlled study

JUSTIFICATION: In the literature one does not find a pharmacological treatment that changes the natural history of Spinocerebellar ataxtia type 3 (SCA3). Patients with this disease invariably become dependent.

OBJECTIVES I. To determine safety and tolerability of phenylbutyrate in patients with SCA3.

II. To provide early subsidies on the efficacy of phenylbutyrate in SCA3.

DURATION: 12 months of a double-blind study.

PLACE OF REALIZATION: Hospital de Clínicas de Porto Alegre, Brazil.

NUMBER OF PATIENTS: 20 patients.

CONCOMITANT MEDICATIONS: There are no concomitant medications that are prohibited unless they affect safety parameters of this study (hemogram and platelets; fasting serum glucose, AST, ALT, Gamma-GT, Bilirubins, Prothrombin time, Creatinine, Urea, Na, K, chlorides and arterial gasometry; electrocardiogram and echocardiogram).

MEDICATIONS UNDER INVESTIGATION: Powdered sodium phenylbutyrate in sachets containing each 3g. At the start of the study, the dose will be 15g/day (five sachets) and may be reduced in case of mild adverse events.

OUTCOMES Primary safety outcome: The number of adverse events, interruptions and dose reductions in the two groups (cases and controls).

Efficacy outcomes: Efficacy outcomes are the following scores in both groups: NESSCA, SARA, Barthel, BDI, and WHOQol.

ELIGIBILITY:
Inclusion Criteria:

1. All patients shall have their molecular diagnosis confirmed and expanded polyglutamine tract (CAG) measures already determined.
2. Patients still able to walk with until 8 years of disease duration, and
3. Patients aged 16 years or over will be invited to participate in the study.

Exclusion Criteria:

1. they show electrocardiogram ou echocardiographic alterations suggestive of heart insufficiency at baseline;
2. their serum creatinine levels are higher than 1.2 mg/dL, with the confirmation of renal insufficiency due to the rate of glomerular filtration;
3. they show a history of hypersensibility to sodium phenylbutyrate, and if
4. they (men and women) do not agree to use a reliable contraceptive method during the entire study period and for three months after its end.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of phenylbutyrate in patients with SCA3 | 6 months - 12 months
  The number of adverse events, interruptions and dose reductions in the two groups (cases and controls).

SECONDARY OUTCOMES:
Efficacy of phenylbutyrate in SCA3 on neurological dysfunction and quality of life | 6 months - 12 months
  Efficacy outcomes are the following scores in both groups: NESSCA, SARA, 9-hole peg board test, BDI, and WHOQol.

CONTACTS AND LOCATIONS:
Overall Officials: Laura B Jardim, PhD, Principal Investigator — Medical Genetics Service of Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil